CLINICAL TRIAL: NCT04187521
Title: Heterogeneity Informed Nutrition Therapy for Gestational Diabetes Mellitus
Acronym: HINT-GDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Camille Elise Powe,M.D., Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019p002395; 74256 (Other Grant/Funding Number: Robert Wood Johnson Foundation)
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; pregnancy; diet; nutrition
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sensitivity defect (Other): Participants defined as having abnormal insulin sensitivity without an absolute defect in insulin secretion.
  Interventions: Other: Meal A; Other: Meal B
- Secretory defect (Other): Participants defined as having abnormal insulin secretion without a defect in insulin sensitivity.
  Interventions: Other: Meal A; Other: Meal B
- Unclassified (Other): Participants who cannot be classified as having abnormal insulin secretion or abnormal insulin sensitivity or who have both abnormal insulin sensitivity and abnormal insulin secretion.
  Interventions: Other: Meal A; Other: Meal B

INTERVENTIONS:
Other: Meal A — A breakfast meal with a specific macronutrient proportions.
Other: Meal B — A breakfast meal with a specific macronutrient proportions.

SUMMARY:
The hypothesis for this study is that women with different physiologic subtypes of gestational diabetes (GDM) (insulin secretion deficit vs. insulin sensitivity deficit) will differ in their glycemic responses to meals with different portions of dietary macronutrients. Investigators will determine GDM subtype based on glucose and insulin levels taken at multiple time points during an oral glucose tolerance test. Participants will consume two meals with different macronutrient content while wearing a continuous glucose monitor which will allow investigators to assess the glycemic response to the meals.

DETAILED DESCRIPTION:
Diabetes mellitus can be classified based on impairments in two different physiologic parameters, insulin secretion and insulin sensitivity. The investigator involved in this trial has previously defined GDM subtypes based on underlying physiology and demonstrated that women with GDM and predominant sensitivity defects have an elevated risk of adverse pregnancy outcomes, while women with predominant secretion defects do not appear to carry the same risk. This supports the idea that not all gestational diabetes is the same. Ideal treatment strategies may differ between GDM subtypes. In this trial, investigators will evaluate the postprandial glycemic response to two test meals with different macronutrient content in different GDM physiologic subtypes. Two test meals with different macronutrient proportions have been designed by research dieticians. Participants will eat test meals at home for breakfast in a randomized order after an overnight fast. Participants will complete food and blood sugar diaries, and will wear a continuous glucose monitor, which will measure postprandial glucose.

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of gestational diabetes

Exclusion Criteria:

* Known diabetes mellitus that preceded pregnancy
* Food allergies to components of the test meals
* Use of medications known to affect glucose tolerance
* Have extensive skin changes or diseases making CGM sensor use problematic
* Demonstrated allergy to CGM adhesive
* Inability to adhere to the swimming and bathing instructions
* Plan to have MRI, CT scan, X Ray or diathermy (heat treatment) during the 7-day CGM study period
* Inability to adhere to Vitamin C guidelines during study period (using more than 500 mg of Vitamin C/day which could interfere with the CGM)
* Use of medications known to affect glucose tolerance
* In the opinion of the principal investigator (PI), demonstrate any other factor likely to limit compliance with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 60 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak blood glucose following test meal (CGM) | 15 mins - 3 hours
  Peak postprandial blood glucose after test meal assessed by continuous glucose monitor

SECONDARY OUTCOMES:
One-hour post prandial blood glucose following test meal (SMBG) | 1 hour
  1 hour postprandial blood glucose after test meal on day 2 and day 3 assessed by glucometer
Glucose area under the curve following test meal (CGM) | 3 hours
  Area under the curve of CGM measured glucose from the start of the test meal to three hours after the test meal is started
Meal taste | 1 hour
  Palatability of the test meals measured using a visual analog scale
Meal satiety | 3 hours
  Satiety following meal measured using a visual analog scale
Meal completion | 1 hour
  Percent of test meal finished assessed by photo of completed meal
Peak blood glucose following lunch on day of test meal (CGM) | 15 mins - 3 hours
  Peak postprandial blood glucose after lunch on days of test meals assessed by CGM
One-hour post prandial blood glucose following lunch on day of test meal (SMBG) | 1 hour
  1 hour postprandial blood glucose after lunch on days of test meals assessed by glucometer
Carbohydrate content of lunch after test meal | 6 hours
  Carbohydrate content (grams) of lunch meal following the test meal
Calorie content of lunch after test meal | 6 hours
  Calorie content of lunch meal following the test meal
Peak blood glucose following dinner on day of test meals (CGM) | 15 mins - 3 hours
  Peak postprandial blood glucose after dinner on day of test meal assessed by CGM
One-hour postprandial blood glucose following dinner on day of test meal (SMBG) | 1 hour
  1 hour postprandial blood glucose after dinner on day of test meal assessed by glucometer
Carbohydrate content of dinner after test meal | 6 hours
  Carbohydrate content (grams) of dinner meal following the test meal
Calorie content of dinner after test meal | 6 hours
  Calorie content of dinner meal following the test meal
Mean blood glucose | 24 hours
  Mean blood glucose on the day of the test meal assessed by CGM
Time in target range | 24 hours
  Length of time at which the patient's BG are within goal range (65-140 mg/dl) on the day of test meal assessed by CGM
Time above target range | 24 hours
  Length of time at which the patient's BG is >140 mg/dl on the day of test meals assessed by CGM
Time below target range | 24 hours
  Length of time at which the patient's BG is <65 mg/dl on the day of test meals assessed by CGM
Total caloric intake on the days of test meals | 24 hours
  Total calorie intake on the day that the test meal is consumed

CONTACTS AND LOCATIONS:
Overall Officials: Camille E Powe, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Powe CE, Allard C, Battista MC, Doyon M, Bouchard L, Ecker JL, Perron P, Florez JC, Thadhani R, Hivert MF. Heterogeneous Contribution of Insulin Sensitivity and Secretion Defects to Gestational Diabetes Mellitus. Diabetes Care. 2016 Jun;39(6):1052-5. doi: 10.2337/dc15-2672. Epub 2016 May 13. PMID 27208340